CLINICAL TRIAL: NCT04850391
Title: Interaction of Sleep, Diurnal Eating Pattern, Gut Microbiota, and Obesity
Acronym: ObeApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Helsinki (Other); University of Turku (Other)
Responsible Party: Principal Investigator, Tarja Saaresranta, Principal Investigator, Turku University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ObeApp
Record Dates: First submitted 2021-04-09; First posted 2021-04-20 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Obesity & Overweight
Keywords: obesity; eating window; time-restricted eating; sleep; glucose balance
MeSH Terms: conditions — Obesity; Overweight; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lean-overweight (Active Comparator): BMI 18.5 - 30 kg/m2
  Interventions: Other: Mobile app
- Obese (Active Comparator): BMI > 30 kg/m2
  Interventions: Other: Mobile app
- Obese OSA (Active Comparator): OSAS patients with BMI > 30 kg/m2
  Interventions: Other: Mobile app

INTERVENTIONS:
Other: Mobile app — To compare changes induced by the movile app intervention among the three study groups

SUMMARY:
The goals of the proposed study are 1) to provide scientific basis for the relationship between subjective sleep quality, diurnal eating pattern, gut microbiome, and obesity, 2) to develop and test a pragmatic, cost-effective new tool to advance lifestyle changes using E-health approach, and 3) to compare differences in subjective sleep quality, diurnal eating pattern and gut microbiome at baseline 4) to compare changes induced by the E-health intervention among the three study groups and participants with different work schedules.

DETAILED DESCRIPTION:
The data are fragmented and studies are focusing on interactions of sleep and obesity, eating pattern and obesity, or gut microbiota and obesity, but not the cross-talk of all these factors in the same individual or population. Therefore, we need a multifactorial approach to get a more deep insight on the obesity and weight regulation. Further, novel cost-effective tools to advance lifestyle changes are needed. Emerging evidence suggests that novel countermeasures, such as modulation of the timing of food intake, may be effective strategies in weight control and prevention of obesity. The goals of the proposed study are 1) to provide scientific basis for the relationship between subjective sleep quality, diurnal eating pattern, gut microbiome, and obesity, 2) to develop and test a pragmatic, cost-effective new tool to advance lifestyle changes using E-health approach, and 3) to compare differences in subjective sleep quality, diurnal eating pattern and gut microbiome at baseline 4) to compare changes induced by the E-health intervention among the three study groups and participants with different work schedules.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling 18 - 65 year old adults
* BMI 18.5 - 30 kg/m2 (n = 40, M:F = 1:1)
* BMI > 30 kg/m2 (n = 40, M:F = 1:1)
* OSAS patients with BMI > 30 kg/m2 using nasal continuous positive airway pressure (CPAP) treatment on an average > 4 h/d (n = 40, M:F = 1:1).

Exclusion Criteria:

* Antimicrobial treatment within 3 months prior the baseline visit
* Inflammatory bowel diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Weight | 2 years
  Changes in weight
Waist/Hip ratio | 2 years
  Changes in Waist/Hip ratio
Change in Blood Pressure | 2 years
  Change in Blood Pressure
GHbA1c | 2 years
  Change in GHbA1c
Gut microbiota | 2 years
  Changes in gut microbiota (species, proportions of different species)
Timing of eating | 2 years
  Change in timing of eating
Subjective sleep quality (Pittsburg Sleep Quality Index) | 2 years
  Changes in subjective sleep quality
Excessive daytime sleepiness (Epworth Sleepiness Scale) | 2 years
  Change in excessive daytime sleepiness
Mood (DEPS questionnaire) | 2 years
  Changes in mood

CONTACTS AND LOCATIONS:
Overall Officials: Tarja Saaresranta, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided